CLINICAL TRIAL: NCT03194516
Title: A Ketogenic Diet Pilot Study for Overweight Prostate Cancer Patients on Active Surveillance
Brief Title: Ketogenic Diet and Prostate Cancer Surveillance Pilot
Acronym: GCC 1717
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00072961
Record Dates: First submitted 2017-04-21; First posted 2017-06-21 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; ketogenic diet; overweight, obese
MeSH Terms: conditions — Prostatic Neoplasms; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surveillance — The investigators propose an 8-week ketogenic diet intervention with pre-/post-intervention assessment of serum and tissue metabolic and inflammatory biomarkers, including metabolomics analysis, among a sample of 12 overweight or obese prostate cancer patients on active surveillance. There will be no randomization; all patients will receive the diet intervention.

SUMMARY:
Men with indolent forms of prostate cancer are managed expectantly using active surveillance, with a goal of delaying treatment and its deleterious side effects. However, almost 50% of men experience progression with this approach and require treatment. Elevated body mass index (BMI) is associated with a dramatically increased risk of progression to higher grade prostate cancer. The goal of the proposed research is to gather preliminary data evaluating the effects of a promising dietary strategy to delay cancer progression in overweight and obese prostate cancer patients undergoing active surveillance. The investigators hypothesize that a ketogenic diet intervention may reduce BMI and favorably alter the prostate microenvironment.

DETAILED DESCRIPTION:
More than 1.6 million new cases of cancer are estimated in the United States in 2016, with almost 600,000 individuals dying from the disease. Prostate cancer alone is responsible for 180,000 new diagnoses per year and remains the most common new cancer diagnosis for men.

Current treatment options for prostate cancer include surgery, radiation, high-intensity focused ultrasound, and cryotherapy. Although typically successful, these strategies carry significant risks for incontinence, erectile dysfunction, and local tissue injury. As a result, for a select subgroup of men with more indolent forms of prostate cancer, active surveillance has become the preferred management strategy. This approach entails periodic laboratory testing, with prostate-specific antigen (PSA) checks at intervals of 3-6 months, and repeat prostate biopsies every 1-2 years or earlier if indicated by PSA elevations. Treatment interventions are typically withheld unless re-biopsy results indicate progression to more aggressive disease. Prospective data comparing surgery and active surveillance have demonstrated improved quality of life outcomes with the latter approach . Not surprisingly, national registry data shows that active surveillance usage has increased from <15% between 1990 and 2009 to >40% between 2010 and 2013 for eligible patients . In order to ensure proper patient selection for active surveillance, MRI guided confirmation biopsies have become standard of care options. Almost one-third of patients will be found to harbor more aggressive cancer than revealed by their initial biopsy. Ideally, treatment could be delayed indefinitely for properly selected patients.

Although surveillance offers a reprieve from cancer treatment and its potential negative sequelae, this benefit appears temporary for many men. Institutional cohort data indicate that 36%-55% of men on active surveillance will require treatment for disease progression within 10 years. One notable risk factor for disease progression during surveillance is overweight and obesity. In a study of 565 prostate cancer patients on surveillance, a 50% increased risk of pathologic progression was associated with every 5 kg/m2 increase in BMI over 25. These results support additional evidence linking weight gain with an increased risk of prostate cancer recurrence after surgery. They have also prompted studies examining pre-surgical weight loss using caloric restriction to mitigate the risk associated with obesity. A low carbohydrate, ketogenic approach has been previously studied in small samples of patients with other types of cancer and also proposed for prostate cancer patients.

In brief, a ketogenic diet is a high-fat, low-carbohydrate diet that mimics the metabolic state of long-term fasting. Ketone bodies are generated mainly by ketogenesis in the mitochondrial matrix of liver cells and are subsequently exported via the blood to other organs to cover the energy demands of cells throughout the body. Ketogenic deaminated amino acids such as leucine also feed the citric acid cycle to form ketone bodies. Utilization of a ketogenic diet as an adjuvant prostate cancer therapy is particularly intriguing given recent preclinical data demonstrating that ketones function as endogenous histone deacetylase (HDAC) inhibitors. HDAC inhibitors have been shown to inhibit prostate cancer proliferation in preclinical models, and are already being studied in clinical trials. Therefore, the ketogenic diet may have a direct impact on disease progression that may extend beyond the BMI reduction achievable by caloric restriction, exercise or other weight loss strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male Adults ≥ 18 years of age
* New biopsy proven prostate adenocarcinoma meeting NCCN guidelines for active surveillance OR previously diagnosed prostate cancer patients on active surveillance
* Eastern Cancer Oncology Group performance status ≤2
* Life expectancy > 1 year
* BMI ≥ 25 kg/m2

Exclusion Criteria:

* Diabetes mellitus on diabetes medication or insulin therapy
* Prior completion of MRI guided confirmation prostate biopsy
* Use of hormonal therapy including finasteride in the past 6 months
* Concomitant use of oral glucocorticosteroids
* Cholecystectomy within 1 year prior to study entry
* Symptoms requiring immediate surgical intervention or radiation therapy
* Active malignancy other than prostate cancer requiring therapy other than non-melanomatous skin cancers
* Participation in any clinical research study evaluating an investigational drug or therapy within one month prior to enrollment
* Any condition that in the judgment of the investigators would interfere with the subject's ability to comply with the study procedures, tolerate the dietary protocol or interfere with the evaluation of responses
* Unable or unwilling to provide informed consent
* Must not be a female of any age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, community care clinic
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Weight loss | 8 weeks

SECONDARY OUTCOMES:
Changes in Testosterone Level | 8 weeks
Changes in Estrogen Level | 8 weeks
Changes in TNF-Alpha Level | 8 weeks
Changes in C-Reactive Protein Level | 8 weeks
Changes in PSA Level | 8 weeks
Changes in High Density Lipoprotein (HDL) | 8 weeks
Changes in Low Density Lipoprotein (LDL) | 8 weeks
Changes in Triglyceride Level | 8 weeks
Changes in Total Cholesterol Level | 8 weeks
Changes in Fasting Glucose Level | 8 weeks
Changes in Leptin Level | 8 weeks
Changes in Fasting Insulin Level | 8 weeks
Changes in Prostate Tissue Metabolomic Profile | 8 weeks
Changes in Prostate Tissue DNA Methylation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Kaiser, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Maryland GCCC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No